CLINICAL TRIAL: NCT04470440
Title: Thyroid Biological Toxicity and Tumor Response in Patients Treated With NIVOLUMAB 2nd Line in Non-small Cell Bronchopulmonary Cancer
Brief Title: Thyroid Dysfunction and Nivolumab Reponse in NSCLC
Acronym: THYRONIVO
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: THYRONIVO (29BRC19.0228)
Record Dates: First submitted 2020-07-07; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Non Small Cell Lung Cancer Metastatic; Treatment Adverse Effect; Thyroid Dysfunction; Immune Checkpoint Inhibitor; Prognosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, retrospective and monocentric study, conducted at the university Hospital of Brest The primary objective is to assess the association between the occurrence of thyroid dysfunction in patients treated with Nivolumab® for a non-small cell lung cancer and prognosis and therapeutic response The second objective is to assess prognosis and therapeutic response according to severity and subtype of thyroid dysfunction

DETAILED DESCRIPTION:
Cohort characteristics

The patients' characteristics were collected from medicals records: age, gender, smoking status (absent, current or weaned), WHO performance index, neoplastic characteristics (tumor histology, history of brain metastasis, prior radiotherapy treatment, prior therapy lines (defined by the number of chemotherapy or immunotherapy regimens used before Nivolumab® treatment) We also recorded data about expression of tumor PD-L1, LDH levels and the lymphocyte to neutrophil ratio (dNLR) summarized in the LIPI score (Lung immune prognostic index), which distinguishes three categories: good prognosis (normal LDH, dNLR <3), intermediate prognosis (abnormal LDH or dNLR> 3), poor prognosis (abnormal LDH and dNLR> 3),

Treatment schedule and morphological monitoring

Nivolumab® (3mg/kg mg) was administered as an IV infusion for 30 minutes every 2 weeks until disease progression, unacceptable toxicity, or death. Tumor assessment was performed every 2 months until disease progression. Tumor assessment was based on the results of the computerized tomodensitometry (CT) + injection of a radioiodine contrast agent and/or 18F-fluorodeoxyglucose (FDG) positron emission tomography (PET/CT) (18FDG-PET/CT), according to the RECIST 1.1 or iRECIST 1.1 ((immune) Response Evaluation Criteria in Solid Tumors) criterion. In case of a dissociated response (response of a lesion associated with a progression of another lesion) or in case of suspicion of pseudo-progression (increase in size or appearance of new lesions linked to the influx of immune cells within the tumor), a new morphological evaluation after two additional cycles was taken into account.

Thyroid function screening and classification of thyroid dysfunction

Thyroid function screening was performed before (<3 months) and during treatment with Nivolumab® (TSH, free T4 (fT4), free T3 (fT3) ± Anti-thyroid peroxidase antibodies (TPOAb) and/or TSH receptor antibodies (TRAbs) were measured by electrochemiluminescence (Reference laboratory values were: TSH, 0.27-4.20 mIU/L; fT4, 11.6-22.0 pmol/L; fT3, 4.0-6.8 pmol/L; TPOAb, <34 kIU/L; and TRAb, <1.75 U/L

For classification of thyroid dysfunction, the CTCAE classification was not taken into account because it is not adapted to thyroid dysfunction that is often asymptomatic. Only abnormalities of the thyroid function tests were considered as follow:

1. Patients with abnormalities of TSH level were classified in the group "Thyroid Dysfunction +" and those with normal TSH level were classified in the group "Thyroid Dysfunction -". In case of normal TSH with isolated abnormality of peripherical hormone fT4 and/or fT3, the patient was classified in the "Thyroid Dysfunction -" group;
2. Depending on the level of peripheral thyroid hormones (i.e. fT3 and fT4): subclinical thyroid dysfunction was defined by an abnormal TSH without abnormality of the peripheral hormones and overt thyroid dysfunction was defined by an abnormal TSH associated with at least one abnormality of the peripheral hormones T3 or T4L;
3. Depending on the TSH level: moderate thyroid dysfunction was defined by a TSH level between 0.1 mIU/L and 0.27 mIU/L or between 4.2 mIU/L and 10 mIU/L, and severe thyroid dysfunction was defined in case of TSH ≤ 0.1 mUI/L or ≥ 10 mUI/L, respectively for hyperthyroidism and hypothyroidism;
4. Depending on the type of thyroid dysfunction, we classified each patient in three categories isolated hypothyroidism, isolated thyrotoxicosis and thyroiditis (thyrotoxicosis then hypothyroidism).

ELIGIBILITY:
Inclusion Criteria:

* patients at least 18 years old and had histologically confirmed locally advanced stage (IIIB) or metastatic (IV) non-small cell lung cancer with disease progression;
* treated with Nivolumab® as second or more therapeutic line
* in the oncologic department university hospital of Brest
* during the inclusion period between July 20, 2015 to June 30, 2018.

Exclusion Criteria:

* patients whose primary tumor was not from bronchopulmonary origin
* patients with a history of total thyroidectomy and/or having previously treated with levothyroxine and/or having a thyroid dysfunction previously to the introduction of Nivolumab®
* patients not having any thyroid monitoring during Nivolumab® treatment, and those for which data were missing
* patients who expressed their opposition to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated with Nivolumab® for a non-small cell lung cancer as a second line
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
overall survival | up to 48 months
  OS was defined as the time between the introduction of Nivolumab® and death

SECONDARY OUTCOMES:
objective response rate (ORR) | up to 48 months
  The ORR was defined as a partial or complete response
disease control rate (DCR) | up to 48 months
  DCR was defined as stability or as an objective response
Progression-free survival | up to 48 months
  PFS is defined as the time between the introduction of Nivolumab® and the date of progression or death.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning trois month and ending five year following the end of the study
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.